CLINICAL TRIAL: NCT02756793
Title: Stereotactic Radiotherapy for Oligo-Progressive Metastatic Cancer (The STOP Trial): A Randomized Phase II Trial
Brief Title: Stereotactic Radiotherapy for Oligo-Progressive Metastatic Cancer (The STOP Trial)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, David Palma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOP
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care Treatment (Active Comparator): Patient treatment may include the following 3 options, at the discretion of the treating physicians:
  * Continue with current systemic agent(s)
  * Observation
  * Switch to next-line treatment
  Interventions: Other: Standard of Care Treatment
- Stereotactic Ablative Radiotherapy (SABR) (Experimental): SABR is delivered to all sites of progressive disease with continuation of current systemic agents. Further oligo-progressive lesions may be treated with SABR if possible. Upon progression at sites not amenable to SABR, the patient may receive any of the options in Arm 1.
  Interventions: Radiation: Stereotactic Ablative Radiotherapy (SABR)

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy (SABR) — Patients will receive stereotactic ablative radiotherapy to all sites of progressive disease, with continuation of current systemic agents.
  Arms: Stereotactic Ablative Radiotherapy (SABR)
Other: Standard of Care Treatment — May include:
  * Continue with current systemic agent(s)
  * Observation
  * Switch to next-line treatment
  Palliative radiotherapy is allowed in this arm.
  Arms: Standard of Care Treatment

SUMMARY:
A multicenter randomized phase II trial of stereotactic body radiotherapy for oligo-progressive metastatic cancers. Eligible patients will be randomized in a 1:2 ratio between receiving their standard of care therapy or stereotactic ablative radiotherapy (SABR) to all sites of oligo-progressive lesions.Radiotherapy will be administered as soon as possible following randomization, and subjects will be followed until next disease progression. The primary outcome is progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Willing to provide informed consent
* Histologically confirmed Non-Small Cell Lung Cancer (NSCLC) with metastatic disease detected on imaging. Biopsy of metastasis at some time point prior to enrollment is preferred, but not required.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy > 3 months
* Patient has received treatment with systemic therapy (either cytotoxic or targeted, including maintenance therapies) during the past 6 weeks. This most recent systemic therapy agent must have been delivered for a total of at least 3 months, with an initial partial response (PR), complete response (CR) or stable disease (CR) prior to the development of oligo-progressive lesions.
* Oligoprogression, defined as Response Evaluation Criteria in Solid Tumors (RECIST)-documented progression in up to 5 individual lesions, with no previous radiation or radiofrequency ablation to those sites. Oligoprogression may be defined as:
* Progression of an individual metastasis according to RECIST 1.1 criteria
* Unambiguous development of a new metastatic lesion at least 5mm in size
* Progressive enlargement of a known metastasis on 2 consecutive imaging studies 2- 3 months apart with a minimum 5mm increase in size from baseline
* All sites of oligoprogression can be safely treated
* Maximum 3 progressing metastases in any single organ system (i.e. lung, liver, brain, bone), and the total number of metastases must be 5 or less

Note for Patients with Brain Metastases: For patients with brain metastases and oligo-progression elsewhere where stereotactic radiation to the brain is deemed to be warranted, this must be specified prior to randomization. If randomized to Standard Arm, patient would receive stereotactic radiation to brain only. If randomized to Experimental Arm, patient would receive stereotactic radiation to brain and to body lesions

Exclusion Criteria:

* Serious medical comorbidities precluding radiotherapy, such as ataxia-telangiectasia or scleroderma. For patients with oligoprogressive lesions in the lung or thorax, this includes interstitial lung disease
* Prior radiotherapy to a site requiring treatment
* Malignant pleural effusion
* Inability to treat all sites of enlarging, oligoprogressive disease
* Clinical or radiological evidence of spinal cord compression or tumor within 3mm of spinal cord on MRI
* Any other condition which in the judgment of the investigator would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-10; Primary Completion 2022-07-31 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 5 years
  Progression-Free Survival is defined as the time from randomization to progression of disease or death from any cause

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Overall survival is defined as they time from randomization to death from any cause
Quality of Life | 5 years
  Quality of life in domains of physical, social/family, emotional, and functional well-being will be assessed with the Functional Assessment of Cancer Therapy (FACT-G)
Toxicity | 5 years
  Toxicity related to radiation treatment will be assessed by the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4 for each organ treated (i.e. liver, lung, bone)
Lesional Control Rate | 5 years
  Local control rate of lesions treated with SABR
Total Time on Chemotherapy | 5 years
  Duration of systemic therapy treatment
Duration of current systemic agent treatment after SABR | 5 years
  Arm 2 only
Location of sites of further progression after SABR | 5 years
  Sites of progressive disease after SABR are captured in follow up

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - Alberta Health Services-Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer - Prince George, Prince George, British Columbia
  - BC Cancer Fraser Valley Centre, Surrey, British Columbia
  - BC Cancer Agency Branch, Vancouver, British Columbia
  - BC Cancer - Victoria Centre, Victoria, British Columbia
  - London Regional Cancer Program, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schellenberg D, Gabos Z, Duimering A, Debenham B, Fairchild A, Huang F, Rowe LS, Severin D, Giuliani ME, Bezjak A, Lok BH, Raman S, Chung P, Zhao Y, Ho CK, Lock M, Louie AV, Lefresne S, Carolan H, Liu M, Yau V, Ye A, Olson RA, Mou B, Mohamed IG, Petrik DW, Dosani M, Pai H, Valev B, Gaede S, Warner A, Palma DA. Stereotactic Ablative Radiation for Oligoprogressive Cancers: Results of the Randomized Phase 2 STOP Trial. Int J Radiat Oncol Biol Phys. 2025 Jan 1;121(1):28-38. doi: 10.1016/j.ijrobp.2024.08.031. Epub 2024 Aug 19. PMID 39168356
- [Derived] Lee J, Koom WS, Byun HK, Yang G, Kim MS, Park EJ, Ahn JB, Beom SH, Kim HS, Shin SJ, Kim K, Chang JS. Metastasis-Directed Radiotherapy for Oligoprogressive or Oligopersistent Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2022 Jun;21(2):e78-e86. doi: 10.1016/j.clcc.2021.10.009. Epub 2021 Nov 18. PMID 34903471